CLINICAL TRIAL: NCT03733886
Title: A Randomised Sham-controlled Double-blinded Study of Burst Spinal Cord Stimulation for Chronic Peripheral Neuropathic Pain.
Brief Title: Burst Spinal Cord Stimulation for Neuropathic Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Bård Lundeland, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017/402/REK nord
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Peripheral Neuropathic Pain; Radiculopathy; Lower Back Pain
MeSH Terms: conditions — Radiculopathy; Low Back Pain

STUDY DESIGN:
Intervention Model Description: N-of-1-study.
  Each patient will go through three treatment cycles each consisting of two weeks of active treatment and two weeks of sham in randomised order. In total the study period will be 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Burst SCS (Active Comparator): In the active comparator the burst SCS system will be turned on according to randomisation.
  A treatment period is a 2-week period where the patient receives either active treatment or sham. Each patient will go through 6 treatment periods (in total 12 weeks). A treatment cycle is a 4-week period with two treatment periods, one of active treatment and one of sham. Each patient will go through three treatment cycles.
  Interventions: Device: Burst SCS (Abbott Proclaim IPG and single lead Abbott Octrode at level Th9/10)
- Sham (Sham Comparator): In the sham comparator the burst SCS system will be turned off according to randomisation.
  Interventions: Device: Burst SCS (Abbott Proclaim IPG and single lead Abbott Octrode at level Th9/10)

INTERVENTIONS:
Device: Burst SCS (Abbott Proclaim IPG and single lead Abbott Octrode at level Th9/10) — Burst SCS implies high frequency SCS treatment in intermittent packets with stimulation below detection level. Abbott BurstDR at default setting: Pulse width 1000 microseconds, frequency 500 Hz/40 Hz, continuous stimulation (no cycling). Pulse amplitude at maximum 60% of sensory threshold

SUMMARY:
This study will evaluate the effect of Burst spinal cord stimulation (SCS) in the treatment of painful radiculopathy in lower extremity(ies) with or without lower back pain. It is a multicenter double-blinded "n-of-1" RCT with repeated two-week periods of Burst SCS or sham in randomised order.

DETAILED DESCRIPTION:
SCS is a treatment offered to patients with peripheral neuropathic pain, and involves electrical stimulation of the spinal cord. The analgesic effect is possibly mediated via both spinal and supra-spinal mechanisms.

Traditional "tonic" SCS causes paresthesia during treatment, but the newer burst technique (five electrical pulses at 500Hz delivered in intermittent packets of 40 Hz) can be performed below detection level. Thus, it is possible to do double-blinded sham-controlled studies.

In this study, we will study the effect of burst SCS compared with sham on pain intensity and function (Patient-Specific Functional Scale). In addition, we will use several questionnaires (psychometric data, health-related quality of life, sleep, global impression of change, use of analgesics, blinding).

ELIGIBILITY:
Inclusion Criteria:

* History, symptoms and clinical findings consistent with painful radiculopathy in lower extremity(ies) ("probable" or "definite") for at least 3 months, with or without lower back pain. The pain in the extremity(ies) must dominate.
* Understand Norwegian or Swedish language (written and spoken).
* Usual pain intensity ≥ 3.5 / 10 (NRS 0-10)

Exclusion Criteria:

Absolute

* Opioid dose > 100 mg morphine equivalents / day
* Ongoing litigation
* Mental / psychiatric disorder that may affect treatment
* Chronic generalized pain
* Pregnancy
* Hypersensitivity to local anesthetics
* Serious or unclear medical condition such as angina pectoris, severe vascular disorder, infection, malignancy disease, bleeding disorders
* Laminectomy in or above level for planned epidural access
* Spine surgery the last 3 months

Relative

* Ongoing medication that affects coagulation or platelet function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Usual pain intensity in lower extremity(ies) | Will be measured at day 7 to day 13 in each period (to avoid carry-over effects from previous treatment period)
  Numeric rating scale (0-10); usual pain intensity over the last 24 h (day 7-13) with anchor points 0 = No pain and 10 = Worst imaginable pain.

SECONDARY OUTCOMES:
Highest pain intensity in lower extremity(ies) | Will be measured at day 7 to day 13 in each period (to avoid carry-over effects from previous treatment period)
  Numeric rating scale (0-10); highest pain intensity over the last 24 h (day 7-13) with anchor points 0 = No pain and 10 = Worst imaginable pain
Lowest pain intensity in lower extremity(ies) | Time Frame: Will be measured at day 7 to day 13 in each period (to avoid carry-over effects from previous treatment period)
  Numeric rating scale (0-10); lowest pain intensity over the last 24 h (day 7-13) with anchor points 0 = No pain and 10 = Worst imaginable pain
Pain intensity in lower extremity(ies)"now" | Time Frame: Will be measured at day 7 to day 13 in each period (to avoid carry-over effects from previous treatment period)
  Numeric rating scale (0-10); evening pain intensity (day 7-13), with anchor points 0 = No pain and 10 = Worst imaginable pain
Pain unpleasantness | Time Frame: Will be measured at day 7 to day 13 in each period (to avoid carry-over effects from previous treatment period)
  Numeric rating scale (0-10) of pain unpleasantness the last 24 hours, with anchor points 0 = no unpleasantness to 10 = worst imaginable unpleasantness.
Three individually chosen functions that are inhibited by the pain | Time Frame: Will be measured at day 7 to day 13 in each 14-day treatment period (to avoid carry-over effects from previous treatment period)
  The Patient-Specific Functional Scale (Numeric Rating Scale (0-10)) (day 7-13). Anchor points 0 = Unable to perform activity to 10 = Able to perform activity.
Insomnia | Time Frame: Will be measured at the end of each 14-day treatment period
  Insomnia Severity Index questionnaire. (Likert scale: 0= no problem, 4 = very severe problem, total score up to 28. Total score (continuous variable)
EQ-5D index values | Time Frame: Will be measured at the end of each 14-day treatment period
  EQ5D index values according to the EQ-5D UK Time Trade-off (TTO) value set.
EQ-5D self-rated health | Time Frame: Will be measured at the end of each 14-day treatment period
  VAS 0-100 scale.
Patient impression of change | Time Frame: Will be measured at the end of each 14-day treatment period
  Patient Global Impression of Change questionnaire. Patient's global impression of change (function, symptoms and quality of life) since last control (about 14 days prior): Very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse.
Patient blinding questionnaire | Time Frame: Will be measured at the end of each 14-day treatment period
  Does the patient think that the system has been turned on or off
Synptoms of anxiety and depression | Time Frame: Will be measured at the end of each 14-day treatment period
  Hopkins Symptom Checklist-25. Likert scale, from 1(Not at all) to 4 (Extremely), mean of sumscore, 25 in total. Change in totalscore (Continious variable).
Usual pain intensity in lower back | Will be measured at day 7 to day 13 in each period (to avoid carry-over effects from previous treatment period)
  Numeric rating scale (0-10); usual pain intensity over the last 24 h (day 7-13) with anchor points 0 = No pain and 10 = Worst imaginable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Bård Lundeland, PhD, Principal Investigator — Department of Pain Management and Research, Oslo University Hospital
Locations (2):
- Oslo University Hospital, Department of Pain Management and Research, Oslo, Norway
- Uppsala University Hospital, Multidisciplinary Pain Center, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data collected during the trial will be available to other researchers who provide a methodologically sound proposal, and who fulfill institutional guidelines.
Supporting Information: CSR
Time Frame: All of the individual participant data collected during the trial will be available after deidentification, beginning 9 months and lasting 5 years after publication.
Access Criteria: Applications must fulfill institutional guidelines and requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473